CLINICAL TRIAL: NCT01031823
Title: The Multi-media Social Skills Project: Validation of an Intervention for Adolescents With Autism Spectrum Disorders
Brief Title: Adolescent Social Skills Training Program
Acronym: ASST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Michael Murray, Principal Investigator, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 32300
Record Dates: First submitted 2009-12-12; First posted 2009-12-15 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Asperger's Disorder; High-functioning Autism
Keywords: Autism Spectrum Disorder
MeSH Terms: conditions — Asperger Syndrome; Autism Spectrum Disorder

ARMS (1):
- Social Skills Training (Experimental): All participants will take part in this arm of the study.
  Interventions: Behavioral: Multi-Media Social Skills Training Program

INTERVENTIONS:
Behavioral: Multi-Media Social Skills Training Program — All individuals will participate in a twelve week social skills training program designed to enhance the social skills of adolescents with Asperger's Disorder or high-functioning autism. The intervention is comprised of both group therapy and peer generalization.

SUMMARY:
This study is a pre-test, post-test single group design with follow-up at month three. Twenty-four individuals total will participate in this study with 6 participants in each of 4 cohorts. Participants and their parents will complete pre-test measures including both paper and pencil measures and a video-recording to assess the participant's social interaction skills and fluency. These adolescents will participate in both group therapy and peer generalization sessions once a week over the course of twelve weeks. Upon completion of the intervention, participants and parents will complete paper and pencil and video post-test measures. Participants will be encouraged to participate in one follow-up session where the paper and pencil and video measures will be completed again.

DETAILED DESCRIPTION:
After consent , has been obtained, parents will complete the Autism Disorders Interview-Revised (ADI-R; Rutter & LeCourteur, 1995) to determine eligibility and the Checklist for Autism Spectrum Disorder (Mayes & Calhoun, 1999), the Social Responsiveness Scale (SRS; Constantino, 2002), and the Strengths and Difficulties Questionnaire (SDQ; Goodman, 1997) at the initial appointment with the study coordinator.

After assent has been obtained, adolescents will complete the Kaufman Brief Intelligence Test, Second Edition (KBIT-2; Kaufman & Kaufman, 1990) to determine eligibility and the Checklist for Autism Spectrum Disorder (Mayes & Calhoun, 1999), the Strengths and Difficulties Questionnaire (SDQ; Goodman, 1997) and the Loneliness Scale (Asher & Wheeler, 1985). Adolescents will also complete a standardized joint attention assessment.

After the completion of the eligibility and pre-test interventions there will be a wash of participants who do not meet eligibility requirements.

One week before the start of the program, participants will attend an introduction session to the program. At this time, participants will be filmed in a brief interaction with a typically developing peer that will be used as a baseline indicator of their social fluency.

Participants will attend the social skills intervention program once a week for twelve weeks. Each week there will be approximately 90 minutes of group therapy which will be conducted like a seminar class: the principal investigator will teach and review social interaction skills and nuances, participants will be encouraged to take an active role in the class.

During the twelve week intervention there will be three review/fluency building sessions: week four, week eight, and week twelve. The group therapy sessions for these review weeks will simply review the material that was covered during the prior three weeks. Participants will then practice what they have learned by having a conversation with a peer that will be taped.

Following the group therapy session each week, participants will join six typically developing peers in a 90 minute introductory photography class taught by one of the study's co-investigators. The photography class will give the participants the opportunity to practice the skills learned in group therapy with their peer group.

Participants will once again complete a battery of clinical and self-report outcome measures which will serve as the post-test measurements for the study. They will be filmed in a brief interaction with a typically developing peer which will be coded to obtain post-test social interaction skills and fluency scores. These evaluations will occur at completion of social skills program, and at three month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Between 13 and 17 years of age
* A primary diagnosis of Asperger's Syndrome or high-functioning autism, as confirmed by the Autism Disorders Interview-Revised (ADIR; Rutter & LeCourteur, 1995)
* An IQ of 70 or above on the Kaufman Brief Intelligence Test, Second Edition (KBIT-2; Kaufman & Kaufman, 1990)
* Local to Central Pennsylvania region

Exclusion Criteria:

* A significant language delay
* Difficulty with aggression directed at peers
* A primary thought disorder
* A secondary disorder of anxiety or depression so severe as to prevent the individual's participation in the treatment

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2013-07-10 (Actual)

PRIMARY OUTCOMES:
Social Fluency | 12 week, 3 month

SECONDARY OUTCOMES:
Loneliness Scale (Asher & Wheeler, 1985) | 12 week, 3 month
Social Responsiveness Scale (SRS; Constantino, 2002) | 12 week, 3 month
Strengths and Difficulties Questionnaire (SDQ; Goodman, 1997) | 12 week, 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Micheal J Murray, M.D., Principal Investigator — Penn State College of Medicine, Penn State Milton S. Hershey Medical Center
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States